CLINICAL TRIAL: NCT03359499
Title: Impact of Bacillus Clausii Administration on Irritable Bowel Syndrome Patients - a Pilot Study
Brief Title: Impact of Bacillus Clausii Administration on Irritable Bowel Syndrome Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Britanico (Other)
Responsible Party: Principal Investigator, Juan Sebastian Lasa, Clinical Professor, Hospital Britanico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB744
Record Dates: First submitted 2017-11-25; First posted 2017-12-02 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — clausin peptide, Bacillus clausii; Nutrition Assessment; Trimebutine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacillus clausii (Experimental): Bacillus clausii administered orally for two weeks plus standard dietary advice for non-constipated irritable bowel syndrome
  Interventions: Drug: Bacillus clausii
- Antispasmodic (Other): Trimebutine administered orally for two weeks plus standard dietary advice for non-constipated irritable bowel syndrome
  Interventions: Drug: Trimebutine

INTERVENTIONS:
Drug: Bacillus clausii — Oral suspension administered BID
  Other Names: Dietary advice
  Arms: Bacillus clausii
Drug: Trimebutine — One tablet of 200 mg of trimebutine administered BID
  Arms: Antispasmodic

SUMMARY:
Probiotics have been proposed as useful therapeutic alternatives for the treatment of irritable bowel syndrome patients. Bacillus clausii is a probiotic that has been used for the treatment of acute diarrhea among adults and pediatric patients, as well as an adjunctive therapy for the treatment for Helicobacter pylori infection. It has been proposed that Bacillus clausii is effective for the treatment of irritable bowel syndrome-related symptoms (especially diarrhea and bloating) in non-controlled trials. The aim of the proposed investigation is to determine whether the administration of Bacillus clausii during two weeks plus dietary advice compared to antispasmodics plus dietary advice would be an effective and safe alternative.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with non-constipated irritable bowel syndrome according to Rome IV criteria

Exclusion Criteria:

* Allergy to Bacillus clausii spores
* Prior treatment with antibiotics or probiotics (4 weeks)
* Not willing to fulfill symptom diary
* Pregnancy or breastfeeding
* Clinical suspicion of organic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-08-12 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Symptomatic response | After two weeks of treatment
  Decrease of at least 50% of symptom severity score - The Irritable Bowel Syndrome Symptom Severity Scale, which consists of five visual analogue scale- questions: their values range from 0 to 100, thus the total score ranges from 0 to 500. Based on previously published studies, clinical response will be defined as a decrease in at least 50% of the initial score

SECONDARY OUTCOMES:
Symptomatic relapse | Four weeks after treatment completion
  An increase of at least 30% in the symptomatic score based on daily follow up. The score that will be used is the The Irritable Bowel Syndrome Symptom Severity Scale, which consists of five visual analogue scale- questions: their values range from 0 to 100, thus the total score ranges from 0 to 500.

CONTACTS AND LOCATIONS:
Overall Officials: Juan S Lasa, MD, Principal Investigator — Hospital Britanico
Locations (1):
- Hospital Britanico, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided